CLINICAL TRIAL: NCT00048490
Title: Drug-Refractory Neocortical Epilepsy: rTMS Treatment
Brief Title: Transcranial Magnetic Stimulation to Treat Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030024; 03-N-0024
Record Dates: First submitted 2002-10-31; First posted 2002-11-01 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-10

CONDITIONS: Epilepsy
Keywords: Seizures; Magnetism; Brain; Stimulation; Therapy; Epilepsy
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation (TMS)

SUMMARY:
This study will use transcranial magnetic stimulation, or TMS (described below), to treat epilepsy in certain patients whose seizures persist despite optimum medical treatment. TMS used in this study is intended to lessen the number of seizures a patient has by decreasing excitability of the brain in the region where the seizures originate.

Patients between 5 and 65 years of age who have had epilepsy for two or more years and have had at least one seizure a week for at least 6 months may be eligible for this 18-week study. Their seizures must come from a neocortical focus-that is, near the surface of the brain. Candidates will be selected from the NIH Epilepsy clinic and will be screened with an electroencephalogram (EEG), magnetic resonance imaging (MRI) scans, and blood tests.

Participants will keep a diary of the seizures they experience over an 8-week period. After the 8 weeks, they will come to the NIH outpatient clinic for 6 consecutive days for the following procedures:

* Day 1: A regular clinic visit, plus 6 hours of video-EEG recording (described below)
* Days 2 through 5: Video-EEG monitoring and TMS as follows:

8:00 - 11: 00 a.m. 3 hours video-EEG monitoring

11:00 - 12:30 p.m. TMS (includes set-up time; actual stimulation time lasts 30 minutes)

12:30 - 3:00 p.m. Lunch + rest

3:00 - 4:30 p.m. TMS

4:30 - 7:30 p.m. 3 hours video-EEG monitoring

(On the fifth day, subjects will have 6 hours of video-EEG monitoring in the afternoon instead of 3 hours.)

Participants will be randomly assigned to one of two TMS groups. One group will have TMS delivered in a way that is thought to have a chance of reducing seizures; the other will have sham, or placebo, stimulation.

When the TMS sessions are completed, participants will keep a diary of their seizures for another 8 weeks.

Transcranial Magnetic Stimulation

For TMS, an insulated wire coil is placed on the subject's scalp. A brief electrical current passes through the coil, creating a magnetic pulse that travels through the scalp and skull and causes small electrical currents in the cortex, or outer part of the brain. The stimulation may cause muscle, hand or arm twitching, or may cause twitches or temporary tingling in the forearm, head, or face muscles. During the stimulation, electrical activity of muscles is recorded with a computer or other recording device, using electrodes attached to the skin with tape. Some TMS sessions may be videotaped.

Video-EEG Recordings

The EEG recording device is housed in a small pouchlike container that is worn below the shoulder, attached to a belt worn around the waist.

DETAILED DESCRIPTION:
In this study, we will use repetitive transcranial magnetic stimulation (rTMS) at 1.0 Hz to treat patients with poorly controlled neocortical epilepsy refractory to pharmacological treatments as a continuation of our previous study (1.0 Hz TMS in 24 patients with refractory partial epilepsy). Previously, we observed that 1.0 Hz rTMS reduced seizure frequency during the first 2 weeks after TMS, although the difference did not reach statistical significance. However, the results suggested that patients with neocortical temporal foci would have a better response than those with mesial temporal foci. We wish to see whether rTMS leads to a significant reduction in seizure frequency in neocortical epilepsy considering the depth of magnetic field. The design will include two parallel groups, one receiving active treatment, and one sham stimulation directed away from the epileptic focus. The patients and the rating physicians will be blinded to the treatment. 1.0 Hz TMS is a rate proven to induce long term depression in animal models and reported to decrease the excitability of both human and animal cerebral cortex. Our preliminary controlled study showed a trend for reduced seizure frequency after 1.0 Hz stimulation. The main outcome measure will be a reduction in seizure frequency over two weeks after stimulation.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients will be selected from the ERB, NINDS, NIH Epilepsy Clinic.

Age 5 to 65 at entry to protocol.

History of localization-related epilepsy for two or more years.

Patients are on a stable anti-convulsant regimen defined as unchanged medicines and dose modifications lower than 20% in the last month. Blood levels of anticonvulsants will be measured at the beginning of the study, prior to stimulation and after the study to assure that the type and dose of medication will remain constant.

Seizures are not completely responsive to medical treatment (1 or more seizures per week for at least 6 months) and patients have continued seizures despite best medical treatment in the past.

The patients have a localized neocortical seizure focus, based on EEG and neuroimaging findings.

EXCLUSION CRITERIA:

Patients will be excluded from this study if they:

1. are pregnant women (tested with urine pregnancy test). The effects of rTMS on pregnancy are unknown.
2. have severe coronary disease.
3. have increased intracranial pressure as expressed by the presence of papilledema.
4. have cardiac pacemakers.
5. take neuroleptic or antidepressant medications.
6. progressive neurologic disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70
Dates: Start 2002-10; Study Completion 2004-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States